CLINICAL TRIAL: NCT00369863
Title: A Randomized, Placebo-Controlled Clinical Trial of Intravitreal Triamcinolone for Refractory Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8126
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2007-02

CONDITIONS: Diabetic Macular Edema
Keywords: Cystoid macular edema; Diabetic macular edema; Hard exudates; Intravitreal triamcinolone; Macular thickness
MeSH Terms: conditions — Macular Edema | interventions — Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone acetonide

SUMMARY:
To determine the efficacy and safety of intravitreal triamcinolone acetonide for refractory diabetic macular edema.

DETAILED DESCRIPTION:
Overall 80% of diabetic patients with low vision are in the nonproliferative stage and the main cause of decreased visual acuity is macular edema.

According to the early treatment diabetic retinopathy study (ETDRS), the treatment of choice for diabetic macular edema (DME) is laser therapy, which may be neither effective nor curative in some patients.There are many cases which are refractory to laser treatment or not suitable candidates for it.

Corticosteroids might have a beneficial effect on DME. They have been used with different doses and routes (periocular,intravitreal,and slow released implants) for a variety of retinal diseases.

Recently, a few prospective randomized studies, concerning the effect of intravitreal triamcinolone acetonide (IVT) on DME have been published. In their two-year results, Gillies et al. concluded that IVT improved vision and reduced macular thickness in eyes with refractory diabetic macular edema. They showed that this beneficial effect persisted for up to 2 years with repeated treatment.

We also conducted a randomized placebo-controlled clinical trial to determine the safety and efficacy of IVT for intractable DME. Besides, we tried to evaluate the effect of this intervention on angiographic findings of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant macular edema(CSME)
* Clinically significant macular edema(CSME)refractory to initial or supplemental macular photocoagulation

Exclusion Criteria:

* Mono-ocular patients
* History of vitrectomy
* Glaucoma or ocular hypertension
* Significant media opacity
* Traction on the macula

Ages: 44 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76
Dates: Start 2002-06; Study Completion 2003-06

PRIMARY OUTCOMES:
Central macular thickness

SECONDARY OUTCOMES:
Visual acuity
intraocular pressure
Cataract progression
Cystoid macular edema
Macular hard exudates
Macular leakage severity in FA

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad - Hossein Dehghan, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Labbafinejad Medical Center, Tehran, Tehran Province, Iran